CLINICAL TRIAL: NCT06191172
Title: The Effect of Person-Centered Care Applied to Patients With Dementia on Nutritional Status
Acronym: Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Kul, MsC, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IstanbulUC-2022/10
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Dementia
Keywords: dementia; person-centered; Edfed; feeding difficulty
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EXPERIMENT I (Experimental): Reminiscence therapy intervention group
  Interventions: Behavioral: Reminiscence Therapy
- EXPERIMENT II (Experimental): Montessori application initiative group
  Interventions: Behavioral: Montessori application
- EXPERIMENT III (Experimental): Environmental initiative group
  Interventions: Behavioral: Environmental Layout
- EXPERIMENT IV (Experimental): Application of contrast ergonomic special equipment initiative group
  Interventions: Behavioral: Application of contrast ergonomic special equipment
- CONTROL GROUP (No Intervention): ORDINARY CARE

INTERVENTIONS:
Behavioral: Reminiscence Therapy — Old objects and pictures of old objects that facilitate remembering about weekly topics will be taken to the institution by the researcher, and individuals within the scope of the research will be asked for their own photographs, if any.
  Arms: EXPERIMENT I
Behavioral: Montessori application — Drill toy Matching puzzle Chickpeas, rice sorting Lock, zipper Counting beans Making a tie Taking and pouring food with a scoop
  Arms: EXPERIMENT II
Behavioral: Environmental Layout — Dining place Music Lighting Heat
  Arms: EXPERIMENT III
Behavioral: Application of contrast ergonomic special equipment — White tablecloth Beveled red blue and yellow blue plate Ergonomic yellow and red fork, spoon and cup
  Arms: EXPERIMENT IV

SUMMARY:
The aim of this study is to examine the effect of person-centered care on nutritional status of patients with dementia.

In this study, we think that since the practices that reduce the eating difficulties of patients with dementia and prevent possible problems will be applied in a person-centered manner, a different perspective will be developed in this field and will affect the care of the patients more positively.

DETAILED DESCRIPTION:
In line with the observations made and the patient's wishes, Montessori application, landscaping, special equipment such as high-contrast colored crockery, flatware, and spill-free containers, positive communication, effectiveness Person-centered care interventions such as activities will be implemented and their effects on nutritional status will be evaluated (Pre-test - post-test).

test randomized control group experimental design). No intervention will be made to the control group, they will only be observed.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years old,
* Being diagnosed with dementia
* Being able to step on the scale (no lower extremity loss)

Exclusion Criteria:

* Acute disease state (pneumonia),
* Patients with PEG,
* Patients with severe visual and hearing impairment,
* Mild dementia patients,
* Parkinson's patients,
* Patients with head trauma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Edfed score | one month
  Change in edfed score after one month of application

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Istanbul, Sıslı, Turkey (Türkiye)